CLINICAL TRIAL: NCT06834776
Title: Evaluation of Neuromuscular Blockade Responses in Statin-Using and Non-Using Patients Undergoing Elective Surgery Under General Anesthesia, Monitored by Train-of-Four (TOF)
Brief Title: Evaluation of Neuromuscular Blockade Responses in Statin-Using and Non-Using Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, Ass. Prof. Dr., Ankara City Hospital Bilkent
Other Study IDs: TABED 1-24-830
Record Dates: First submitted 2025-01-31; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-12

CONDITIONS: Neuromuscular Blockade; Statin-Associated Myopathy; Neuromuscular Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- cohort A: statin-use
  Interventions: Diagnostic Test: TOF (Train-of-Four) monitoring for depth of neuromuscular blockade.
- Cohort B: statin-nonuse
  Interventions: Diagnostic Test: TOF (Train-of-Four) monitoring for depth of neuromuscular blockade.

INTERVENTIONS:
Diagnostic Test: TOF (Train-of-Four) monitoring for depth of neuromuscular blockade. — General anesthesia with propofol and fentanyl induction followed by rocuronium for neuromuscular blockade; maintenance with desflurane and remifentanil.

SUMMARY:
This study aims to compare the neuromuscular blockade responses in patients undergoing elective surgery under general anesthesia, with a focus on the use of statins. The study will assess the depth of neuromuscular blockade, recovery time, and postoperative residual curarization using Train-of-Four (TOF) monitoring, with the primary goal of determining whether statin use alters the neuromuscular blockade management.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* ASA classification I, II, III
* BMI 18-30
* Statin use for at least 3 months or no prior statin use
* Elective surgery requiring general anesthesia with endotracheal intubation
* Signed informed consent for participation in the study

Exclusion Criteria:

* ASA classification IV or higher
* BMI <18 or >30
* History of liver or renal insufficiency (creatinine >1.6, liver function tests >2x normal)
* Neuromuscular, psychiatric, or neurological disorders
* Pregnancy
* Use of drugs affecting neuromuscular function (e.g., anticonvulsants, aminoglycosides)
* History of malignant hyperthermia
* Respiratory disorders, including sleep apnea
* Allergy to anesthetic drugs used in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Statin-Using and Non-Using Patients Undergoing Elective Surgery Under General Anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Time to reach TOF count 0 | 0th minute
  time from administration of rocuronium to reach TOF count 0
Time to reach TOF 40 | about 40th minute
  time to intraoperatively TOF reached 40
Time to reach TOF 90 (reversal of neuromuscular blockade) | about 60th minute
  Measured postoperatively after sugammadex administration and additional doses if required.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Emen, ass. Dr., Study Chair — Ankara City Hospital Bilkent

IPD SHARING:
Plan to Share IPD: Undecided